CLINICAL TRIAL: NCT02159157
Title: A Randomized, Controlled Trial to Determine the Effects of an Exercise Intervention on Physical Activity During Chemotherapy for Patients With Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Mary Chamberlin, Mary Chamberlin, MD, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D12030
Record Dates: First submitted 2014-05-05; First posted 2014-06-09 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Early Stage Breast Cancer
Keywords: breast cancer, exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (No Intervention): Physical Therapy consult for post op care and general physical activity recommendation 1-4 weeks prior to starting chemotherapy.
  Phone calls designed to support the patient to maintain current activity level.
- Arm B (Placebo Comparator): Physical Therapy consult for post-op care 1-4 weeks prior to starting chemotherapy.
  Exercise prescription aimed at increasing physical activity by a minimum of 10 MET hours/week.
  Motivational phone calls aimed at encouraging the patient to adhere to their exercise prescription.
  Interventions: Behavioral: Exercise prescription

INTERVENTIONS:
Behavioral: Exercise prescription — A physical therapist will design an exercise plan for each participant on the intervention arm. The participants randomized to the intervention arm will also receive phone calls to assist with tracking the study participant's exercise and motivating the study participant to adhere to the exercise prescription.
  Arms: Arm B

SUMMARY:
This study is designed to randomly assign breast cancer patients requiring and agreeing to chemotherapy into two groups. One group will be receive an exercise prescription aimed at increasing physical activity by a minimum of 10 MET (metabolic equivalent task) hours per week. The other group will not receive a exercise prescription but their activity will be recorded. The hypothesis is that participants that are most active will exhibit improved chemotherapy completion rates, improved fitness, less fatigue and lower levels of markers for inflammation in their blood.

DETAILED DESCRIPTION:
This is a prospective, randomized, single institution feasibility trial. The efficacy of an exercise intervention during chemotherapy for sedentary breast cancer patients will be tested. The investigators goal is to recruit 120 women and men. Assuming 20% attrition rate, 96 will be randomized to two arms, comparing patients assigned to a physical activity program plus general health education materials versus patients assigned to receive standard general health education materials only. Study measures will be obtained before intervention, at 24 weeks, and at the end of the intervention, approximately week 32.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men with histologically confirmed breast cancer and no evidence of metastatic disease with a recommendation to begin chemotherapy within 4 weeks.
2. Patients must have recovered from prior surgery.
3. Patients must be able to walk unassisted without oxygen
4. Patients must complete the Physical Activity Readiness questionnaire with "No" answers to all questions; if patient responds with YES answers, OR IS OVER AGE 69, approval must be obtained from the patient's Primary care physician or treating medical oncologist to participate in the study.
5. Able to fast for 12 hours for blood work and Basal Metabolic Rate measurement.
6. Karnofsky performance status > or = to 80%.
7. Previous or ongoing Physical therapy treatments are acceptable.
8. Participants may be enrolled on other treatment-based clinical trials but may not be enrolled on any other weight loss trials.
9. Participants must have a baseline activity level of < 150 minutes/wk of moderate to vigorous activity as calculated using the moderate to vigorous components of the LTEQ (leisure time exercise questionnaire) for physical activity (completed during screening).

Exclusion Criteria:

1. Patients less than 18 years of age.
2. Patients with history of acute MI (myocardial infarction) or CVA (cerebral vascular accident) within the last 12 months.
3. Patients who are oxygen dependent.
4. Patients unable to give informed consent indicating they are aware of the investigational nature of this intervention prior to entry into the study.
5. Patients with a Karnofsky performance status of < 80%.
6. Pregnant.
7. Unable to read or write in English.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-06; Primary Completion 2017-03 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in activity as measured by the Activity Log | from baseline to week 32
  A log will be used to record patient's exercise activity and pedometer data on a weekly and monthly basis.

SECONDARY OUTCOMES:
Received Dose Intensity of chemotherapy (RDI) | 32 weeks
  The RDI is calculated by (delivered dose)/(standard dose) x 100. Delivered dose = (actual total dose in mg/m2)/ (total days required to complete the treatment) Standard dose = (recommended total dose) / (total days planned to complete the treatment)
Change from baseline (day -28 to day 1) fatigue as measured by FACIT-F | baseline (Day -28 to 1), week 24, 32 weeks
  Fatigue as measured by the FACIT-F survey
Change from baseline (day -28 to 1) Absolute neutrophil count and hemoglobin | baseline (Day -28 to 1), 32 weeks
Change from Baseline (day -28 to day 1) C-reactive protein | Baseline (day -28 to day 1) and week 32
  levels of C- reactive protein
Change from Baseline (Day -28 to day 1) Fasting insulin | Baseline (day -28 to day 1) and week 32
  Fasting insulin levels measured in blood at baseline (day -28 to day 1) and week 32
Change from Baseline (day -28 to day 1) of Resting metabolic rate (calculated by Respiratory quotient/ resting energy expenditure measured in kcal/day) | baseline (day -28 to day 1) and week 32
Change in Body composition as indicated by % of total body fat, bone density (g/cm2), and T score | baseline (day -28 to day 1) and week 32
Change in Resting heart rate from baseline (day -28 to day 1) | baseline (day -28 to day 1) and week 32
Change in Waist-hip ratio from baseline (day -28 to day 1) | baseline (day -28 to day 1) and week 32
Change in steps recorded from baseline (day -28 to day 1) as measure by Pedometer data | weekly for 32 weeks
  Average steps per week for weeks 1-32
Measures how likely a person is to continue with exercise prescription. | From baseline to Week 32
  How the participant is feeling about the exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Chamberlin, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

DOCUMENTS (1):
  • Informed Consent Form (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT02159157/ICF_000.pdf